CLINICAL TRIAL: NCT04220021
Title: A Single-Center, Open Label Study to Assess the Safety and Tolerability of Metformin in Subjects With C9orf72 Amyotrophic Lateral Sclerosis Over 24 Weeks of Treatment
Brief Title: Safety and Therapeutic Potential of the FDA-approved Drug Metformin for C9orf72 ALS/FTD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: ALS Association (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201800620; UF2019-001 (Other: University of Florida); OCR20620 (Other: UF OnCore); UF2019-001 (Other: UF Protocol ID); CDMRP AL220089 (Other Grant/Funding Number: USAMRAA); AGR DTD 12-20-2022 (Other Grant/Funding Number: ALS Association)
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: C9orf72 Amyotrophic Lateral Sclerosis (ALS); Frontotemporal Dementia
Keywords: ALS; FTD; Lou Gehrigs Disease
MeSH Terms: conditions — Frontotemporal Dementia; Amyotrophic Lateral Sclerosis | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: All participants receive medication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- C9orf72 positive ALS (Experimental): Subjects with C9orf72 positive ALS will be instructed in the use of Metformin and receive the first dose of Metformin under supervision of the investigator during Visit 1, Day 2.
  Subjects will then continue on Metformin per the dose escalation schedule twice daily for 24 weeks.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin is a widely used, well-tolerated drug that has been used for decades as a first-line defense for treating type 2 diabetes. Its safety has been well established. Subjects will begin treatment with Metformin at a dosage of 500mg with an escalation of dosage by 500mg every week to a maximal dosage of 2000mg. Dosing will be twice daily.
  Other Names: Metformin hydrochloride sustained-release (SR)

SUMMARY:
The primary objective is to assess the safety and tolerability of Metformin in subjects with C9orf72 amyotrophic lateral sclerosis administered for 24 weeks. The overall objective is to determine if Metformin is safe in C9orf72 ALS patients and is a potentially viable therapeutic treatment for C9-ALS that reduces repeat-associated non-canonical start codon - in DNA (non-ATG) (RAN) proteins that are produced by the C9orf72 repeat expansion mutation.

DETAILED DESCRIPTION:
The C9orf72 repeat expansion is the most common cause of amyotrophic lateral sclerosis and frontotemporal dementia (C9-ALS/FTD). Metformin, a well-tolerated diabetes drug, blocks a key pathway for expression of toxic proteins produced from the C9orf72 repeat expansion via repeat associated non-canonical start codon - in RNA (non-AUG) (RAN) translation. In mouse model of C9-ALS/FTD, metformin treatment decreases RAN protein levels and improves disease features. This current study is a small-scale clinical trial to assess the safety and potential efficacy of metformin for the treatment of C9-ALS/FTD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have a diagnosis of probable or definite ALS in accordance with the Revisited El-Escorial Criteria.
* Subjects have a likely diagnosis of chromosome 9 open reading frame 72 (C9orf72) positive ALS/FTD.
* Subjects must be currently on an oral diet and able to take foods, pills and liquids by mouth equivalent to a score of 4 or above on the Functional Oral Intake Scale
* Subjects must have no known allergy to barium sulfate or Metformin.
* Subjects or subject's legally authorized representative must be willing and able to complete informed consent/assent and HIPAA authorization.
* Ability to comprehend and be informed of the nature of the study, as assessed by the PI or Co-Investigators.
* Subjects prescribed to take Metformin at or before the time of first dosing. (The study is open to subjects currently taking Metformin or subjects who have taken Metformin in the past).
* Availability to participate for the entire study duration.
* Female subjects of childbearing potential must have a negative urine pregnancy test prior to Videofluoroscopic Swallow Study (VFSS) exam during Visit 1, 3, and 4.

Exclusion Criteria:

* Subjects who score 3 or below on the Functional Oral Intake Scale
* Subjects who do not carry the C9ORF72 hexanucleotide repeat expansion as determined by laboratory analysis.
* Subjects with a history of clinically significant liver disease, renal disease, or any other medical condition judged to be exclusionary by the investigator.
* Subjects who are unwilling to sign informed consent or subjects who for any other reason in the judgment of investigator are unable to complete the study.
* Female subjects who have a positive urine pregnancy test (βhCG) at screening or visit 1, are trying to become pregnant or are breastfeeding.
* Subjects with active cancer within the previous 2 years, except treated basal cell carcinoma of the skin.
* Subjects who have taken any experimental drug within 30 days prior to enrollment or within 5 half-lives of the investigational drug -whichever is the longer period.
* Subjects with known history or presence of moderate or severe renal impairment as defined by an estimated glomerular filtration rate (eGFR) value below 30 mL/min/1.73 m2.
* Subjects with hepatic impairment as defined by baseline elevations of serum aminotransferases greater than 5 times upper limit of normal or evidence of liver dysfunction (e.g., elevated bilirubin).
* Use of potentially hepatotoxic drugs: (e.g., allopurinol, methyldopa, sulfasalazine).
* Subjects with clinically significant abnormal laboratory values in the judgment of the investigator.
* Subject with implanted electrical device (i.e. cardiac pacemaker or a neurostimulator), metal or metallic clip(s) in their body (i.e. an aneurysm clip in the brain) that will be damaged by participation in the MRI portion of the study.
* Anything else that, in the opinion of the investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ranum, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cedarbaum JM, Stambler N, Malta E, Fuller C, Hilt D, Thurmond B, Nakanishi A. The ALSFRS-R: a revised ALS functional rating scale that incorporates assessments of respiratory function. BDNF ALS Study Group (Phase III). J Neurol Sci. 1999 Oct 31;169(1-2):13-21. doi: 10.1016/s0022-510x(99)00210-5. PMID 10540002
- [Background] Crary MA, Mann GD, Groher ME. Initial psychometric assessment of a functional oral intake scale for dysphagia in stroke patients. Arch Phys Med Rehabil. 2005 Aug;86(8):1516-20. doi: 10.1016/j.apmr.2004.11.049. PMID 16084801
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Background] Watanabe H, Atsuta N, Nakamura R, Hirakawa A, Watanabe H, Ito M, Senda J, Katsuno M, Izumi Y, Morita M, Tomiyama H, Taniguchi A, Aiba I, Abe K, Mizoguchi K, Oda M, Kano O, Okamoto K, Kuwabara S, Hasegawa K, Imai T, Aoki M, Tsuji S, Nakano I, Kaji R, Sobue G. Factors affecting longitudinal functional decline and survival in amyotrophic lateral sclerosis patients. Amyotroph Lateral Scler Frontotemporal Degener. 2015 Jun;16(3-4):230-6. doi: 10.3109/21678421.2014.990036. Epub 2014 Dec 30. PMID 25548957
- [Background] Cammack AJ, Atassi N, Hyman T, van den Berg LH, Harms M, Baloh RH, Brown RH, van Es MA, Veldink JH, de Vries BS, Rothstein JD, Drain C, Jockel-Balsarotti J, Malcolm A, Boodram S, Salter A, Wightman N, Yu H, Sherman AV, Esparza TJ, McKenna-Yasek D, Owegi MA, Douthwright C; Alzheimer's Disease Neuroimaging Initiative; McCampbell A, Ferguson T, Cruchaga C, Cudkowicz M, Miller TM. Prospective natural history study of C9orf72 ALS clinical characteristics and biomarkers. Neurology. 2019 Oct 22;93(17):e1605-e1617. doi: 10.1212/WNL.0000000000008359. Epub 2019 Oct 2. PMID 31578300
- [Background] Atassi N, Berry J, Shui A, Zach N, Sherman A, Sinani E, Walker J, Katsovskiy I, Schoenfeld D, Cudkowicz M, Leitner M. The PRO-ACT database: design, initial analyses, and predictive features. Neurology. 2014 Nov 4;83(19):1719-25. doi: 10.1212/WNL.0000000000000951. Epub 2014 Oct 8. PMID 25298304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 1/3/2020 - 8/28/2023 Recruitment location: University of Florida Neurology Clinic
Groups:
- Enrolled Subjects: Subjects who consented to participate in the study.
Period: Overall Study
Arm/Group | Enrolled Subjects
Started | 41
Completed | 23 (Study participants were defined as having "Completed" the study if they started the study medication and completed the ALSFRS-R evaluation at baseline and 24 weeks.)
Not Completed | 18
Not completed — Withdrawal by Subject | 11
Not completed — Physician Decision | 2
Not completed — Non-study related illness | 5

BASELINE CHARACTERISTICS:
Population: Subjects who consented to the study.
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41
ALSFRS-R [Mean (Standard Deviation); unit: units on a scale] — The Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) is a quickly administered (5 minute) ordinal rating scale (ratings 0-4) used to determine subjects' assessment of their capability and independence in 12 functional activities/questions. The score represents the sum of 12 functional domain items where each item is scored from 0 to 4 (Max score 4 = Normal function; Min score is 0 = No ability to perform the task). The total score range is from 0 to 48, with a score of 48 meaning no functional impairment and 0 meaning complete loss of function across all domains. Population: 23 subjects who started the study medication and who completed the ALSFRS-R evaluations at baseline and 24 weeks.
  units on a scale
    number analyzed (Participants) | 23
    (all) | 38.65 (6.51)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Unexpected Treatment-emergent Adverse Events [Safety and Tolerability]
Description: The safety and tolerability of Metformin in participants with C9orf72 ALS currently treated with Metformin will be evaluated by the number of subjects with treatment-emergent adverse events
Time Frame: Baseline through 24 weeks
Population: Forty-one subjects agreed to participate in the study. Twenty-three participants were defined as having "Completed" the study if they started the study medication and completed the ALSFRS-R evaluation at baseline and 24 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Study Completers: Participants were defined as having "Completed" the study if they started the study medication and completed the ALSFRS-R evaluation at baseline and 24 weeks.
- All Participants: Subjects who consented to participate in the study.
Arm/Group | Study Completers | All Participants
Number analyzed (Participants) | 23 | 41
Participants | 0 | 0

2. Primary Outcome: Change in Repeat Associated Non-AUG (RAN) Protein Levels
Description: Assessment of RAN protein levels in cerebrospinal fluid (CSF) samples from participants calculated as the percentage change in polyglycine-proline (GP) levels in ng/ml at study start & end of the study as measured by Meso Scale Discovery (MSD) assays.
Time Frame: Baseline through week 24.
Population: Data from 17 of the 23 subjects were analyzed: 2 samples were excluded because the subjects were not drug compliant; data from 3 subjects were excluded because GP levels were not reliably detected; 1 sample was excluded because CSF was not able to be collected at the 24 week visit.
Measure: Median (Inter-Quartile Range); unit: % change (ng/ml) from study start to end
Groups:
- Study Completers With Reliable CSF MSD Values: Subjects who remained in the study through Week 24, were compliant with the use of metformin, had reliable MSD values, and who had CSF samples collected at baseline and 24 weeks.
Arm/Group | Study Completers With Reliable CSF MSD Values
Number analyzed (Participants) | 17
% change (ng/ml) from study start to end | -27.93 [-43.98 to -1.91]
Statistical Analysis 1: Comparison: Study Completers With Reliable CSF MSD Values; Sign and binomial test with one-tail analysis where the null hypothesis predicts a 50/50 split (p=0.5) for two outcomes; Test type: Superiority — For the sign and binomial test our two outcomes are decreased (success) percentage change in RAN protein levels and increased (failure) percentage change in RAN protein levels; p = 0.0245, Sign test — A priori test for significance is p less than or equal to 0.05; One-tailed sign and binomial test

3. Secondary Outcome: Change in ALS Functional Rating Scale (ALSFRS-R) Score
Description: The Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) is a quickly administered (5 minute) ordinal rating scale (ratings 0-4) used to assess the capability and independence of subjects across 12 functional activities/questions. The score represents the sum of 12 functional domain items where each item is scored from 0 to 4 (Max score for each functional domain is 4 (Normal function); Minimum score for each functional domain = 0 (No ability to perform the task). The total score range is from 0 to 48, with a score of 48 meaning no functional impairment and 0 meaning complete loss of function across all domains. The mean values reported are at each study visit which occurred at baseline and at approximately 6, 12 and 24 weeks. The total number of days between study visits varied due to scheduling issues.
Time Frame: Baseline through Week 24
Population: Twenty three subjects were analyzed as per protocol at baseline, week 6 and week 24. Twenty-two subjects were analyzed at week 12 because the ALSFRS-R was not completed due to coronavirus disease 2019 (COVID-19) travel difficulties at the 12 week time point. Two subjects who were not compliant with the medication throughout the study were excluded in "Metformin compliant study completers" study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Study Completers: Subjects who started the study medication and who completed the ALSFRS-R evaluations at baseline and 24 weeks.
- Metformin Compliant Study Completers: Subjects who completed the ALSFRS-R at baseline and visit 4 and who were compliant with metformin medication throughout the study
Arm/Group | Study Completers | Metformin Compliant Study Completers
Number analyzed (Participants) | 23 | 21
score on a scale
  Baseline | 38.61 (6.73) | 38.57 (7.06)
  Visit 2-approx. 6 wks | 37.74 (6.76) | 37.57 (7.07)
  Visit 3-approx. 12 wks: number analyzed (Participants) | 22 | 20
  Visit 3-approx. 12 wks | 36.30 (6.92) | 36.33 (7.25)
  Visit 4-approx.24 wks | 34.13 (8.35) | 34.48 (8.68)

ADVERSE EVENTS:
Time Frame: From enrollment up to 24 weeks of treatment.
Description: Adverse Events are reported as defined by ClinicalTrials.gov definition.
Groups:
- Enrolled Subjects: Subjects consented to participate in the study
- Study Completers: Study participants were defined as having "Completed" the study if they started the study medication and completed the ALSFRS-R evaluation at baseline and 24 weeks.
Arm/Group | Enrolled Subjects | Study Completers
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/41 | 0/23
Other Adverse Events (participants affected / at risk) | 35/41 | 16/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=41) | Study Completers (N=23)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Gallbladder disease (Hepatobiliary disorders) | 1 (1) | 0 (0) — Emergency gallbladder removal.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=41) | Study Completers (N=23)
Diarrhea (Gastrointestinal disorders) | 16 (21) | 9 (14)
Nausea (Gastrointestinal disorders) | 6 (6) | 3 (3)
Indigestion (Gastrointestinal disorders) | 4 (6) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 10 (20) | 8 (17)
Abrasion (Skin and subcutaneous tissue disorders) | 4 (8) | 3 (7)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 5 (5)
Unintentional Weight Loss (Metabolism and nutrition disorders) | 5 (6) | 4 (5)
Gastrostomy (Surgical and medical procedures) | 4 (4) | 2 (2)
Post Lumbar Puncture Syndrome (Nervous system disorders) | 7 (8) | 4 (5)
Post-procedural Hematoma (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Backache (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3)
Headache (Nervous system disorders) | 3 (4) | 1 (1) — Headaches unrelated to lumbar puncture

LIMITATIONS AND CAVEATS:
Our C9orf72 ALS metformin clinical trial was not placebo-controlled but ALSFRS-R scores were compared to previously published C9orf72 ALS (PMID: 31578300) and all ALS patient (PMID: 25298304) natural history studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT04220021/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT04220021/ICF_001.pdf